CLINICAL TRIAL: NCT03870425
Title: Distribution of Nutrient Derived Amino Acids and Anabolic Effect in Healthy Elderly Individuals
Brief Title: Distribution of Nutrient Derived Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jakob Agergaard, PhD, Postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BBH 140
Record Dates: First submitted 2019-01-18; First posted 2019-03-12 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Muscle Mass; Protein Intake; Diet Modification; Protein Synthesis; Protein Breakdown; Sarcopenia
Keywords: Dietary protein; Sarcopenia; Protein turnover; Muscle protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINCED-SKEWED (Placebo Comparator): Minced meat administered with a skewed protein distribution pattern
  Interventions: Other: Distribution pattern of dietary proteins (minced meat)
- MINCED-EVEN (Experimental): Minced meat administered with an even protein distribution pattern
  Interventions: Other: Distribution pattern of dietary proteins (minced meat)

INTERVENTIONS:
Other: Distribution pattern of dietary proteins (minced meat) — Study effect of an even or skewed distribution pattern of dietary protein

SUMMARY:
The project examines over several days how the distribution pattern of dietary protein stimulate and affect the protein turnover of important proteins in the aging perspective, such as skeletal muscle proteins.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Between 65-80 years of age

Exclusion Criteria:

* BMI above 30
* Smokers
* Vegetarians
* Diabetes or other metabolic diseases
* Medical treatment which affects protein turnover
* Gastro-intestinal diseases, reduced kidney or liver function, or chronic inflammation diseases
* Elevated blood-pressure or signs of atherosclerosis
* More than 5 hours of regular exercise each week

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 3 days
  Myofibrillar FSR measured by deuterated water technique, by which deuterium labeled alanine incorporation into myofibrillar muscle protein synthesis can be measured.
Net protein balance | 10 hours
  Whole body net protein balance measured during 10 hours acute study. Measured by the application of stable amino acid labeled phenylalanine and tyrosine tracers, by which the protein synthesis, phenylalanine oxidation and protein breakdown can be calculated.

SECONDARY OUTCOMES:
D5-phenylalanine incorporation | 3 days
  D5-phenylalanine incorporation into myofibrillar proteins. Dietary meat proteins are intrinsically labeled with D5-phenylalanine
Muscle protein synthesis | 10 hours
  Myofibrillar protein synthesis (%/hour) measured during 10 hours of the acute study. Calculated from the difference in D8-phenylalanine incorporation from the muscle biopsies taken at 2 hours and 12 hours into the stable amino acid tracer infusion.
Protein synthesis | 10 hours
  Whole body protein synthesis (%/hour) measured during acute study, by the use of stabel amino acid tracer technique.
Protein breakdown | 10 hours
  Whole body protein breakdown (%/hour) measured during acute study, by the use of stabel amino acid tracer technique.
Phenylalanine oxidation | 10 hours
  Phenylalanine oxidation measured during acute study
D5-phenylalanine appearance | 12 hours
  Plasma D5-phenylalanine enrichment after intake of D5-phenylalanine intrinsically labelled meat proteins
Signaling pathways in skeletal muscle | 10 hours
  Intracellular signaling pathways related to protein turnover. Measured by Western blotting technique from the muscle tissue biopsies taken at 2 hours and 12 hours into the acute study.
Plasma insulin | 12 hours
  Plasma insulin concentration during acute study

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agergaard J, Justesen TEH, Jespersen SE, Tagmose Thomsen T, Holm L, van Hall G. Even or skewed dietary protein distribution is reflected in the whole-body protein net-balance in healthy older adults: A randomized controlled trial. Clin Nutr. 2023 Jun;42(6):899-908. doi: 10.1016/j.clnu.2023.04.004. Epub 2023 Apr 8. PMID 37086618